CLINICAL TRIAL: NCT05743296
Title: Differences in Brain Activity in the Application of Upper Limb Exercise Tasks Through Virtual Reality in Chronic Stroke Patients
Brief Title: Differences in Brain Activity in the Application of Upper Limb Exercise Tasks Through Virtual Reality
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-10-117
Record Dates: First submitted 2022-12-22; First posted 2023-02-24 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cross-sectional study, no arm: Experimental: Training with the virtual reality program (MOTOCOG)
  Training consists of 26 minutes task-specific training.

SUMMARY:
This study aims to find out the difference in brain activity when performing upper limb exercise tasks through virtual reality-based MOTOCOG equipment for chronic stroke patients.

DETAILED DESCRIPTION:
This study aims to find out the difference in brain activity when performing upper limb exercise tasks through virtual reality-based MOTOCOG equipment for chronic stroke patients. All participants will participate in tasks for upper limb exercise conducted for 26 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 to 80 years
* FMA Upper scores more than 25 and less than 58
* Patients whose lesions do not include stimulation regions
* Patients with stroke with more than 6 months of onset
* K-MMSE scores more than 24
* patients who can Grasp & release

Exclusion Criteria:

* Difficult to communicate due to severe language impairment.
* Accompanied by an existing serious neurogenic disease
* Existing significant psychiatric disorders such as major schizophrenia, bipolar disorder

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Upper Extremity | Baseline
  Measurement of motor function of upper and lower extremities. The minimum and maximum values are 0 and 66, and higher scores mean a better outcome.

SECONDARY OUTCOMES:
Grip and Tip pinch strength test | Baseline
  The test is to measure the maximum isometric strength of hand, forearm, and finger muscles.
Box & Block Test | Baseline
  The test is used to measure the gross manual dexterity of a patient, or of a person using an upper limb prosthetic device.
9-hole pegboard test | Baseline
  The test is a standardized, quantitative assessment used to measure finger dexterity of a patient.
Jebsen-Taylor Hand Function test | Baseline
  This test is a standardized and objective measure of fine and gross motor hand function using simulated activities of daily living (ADL).

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim J, Kim E, Lee SH, Lee G, Kim YH. Use of cortical hemodynamic responses in digital therapeutics for upper limb rehabilitation in patients with stroke. J Neuroeng Rehabil. 2024 Jul 10;21(1):115. doi: 10.1186/s12984-024-01404-y. PMID 38987817